CLINICAL TRIAL: NCT01873755
Title: Addressing Barriers to Physical Activity in Inner-City Schoolchildren With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-443; 5K23HD065742 (NIH)
Record Dates: First submitted 2013-06-04; First posted 2013-06-10 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Asthma; Children; Physical Activity
Keywords: asthma; children; physical activity; school
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- asthma physical activity intervention (Experimental): two schools will receive intervention
  Interventions: Behavioral: asthma physical activity intervention

INTERVENTIONS:
Behavioral: asthma physical activity intervention — School- and community-based intervention includes several components: a classroom-based physical activity program, asthma awareness week at the school, asthma education for parents and students enrolled in the study, collaboration with child's physician to ensure proper medical treatment of child's asthma asthma education for school personnel

SUMMARY:
This proposal will address the existent gaps in the literature by identifying barriers and facilitators to participation in physical activity in inner-city minority elementary schoolchildren with asthma, more that half of whom are also overweight; developing and refining a school-based intervention in partnership with the community to improve physical activity; and conducting a pilot randomized controlled trial of the intervention to determine feasibility and obtain preliminary data for a future large-scale trial.

DETAILED DESCRIPTION:
Four schools have been recruited for pilot wait-listed cluster randomized clinical trial to determine feasibility for a large-scaled trial. Community-based participatory research approach was utilized to develop an intervention that will be delivered to two schools. Two control schools will receive intervention during year 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* children with active asthma attending 2nd-4th grades in Bronx

Exclusion Criteria:

* other medical conditions preventing participation in physical activity

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2014-05-28 (Actual); Study Completion 2014-06-20 (Actual)

PRIMARY OUTCOMES:
change in physical activity levels | baseline, 6, 9, 12 months follow-up
  physical activity levels will be measured with accelerometers

SECONDARY OUTCOMES:
change in Body Mass Index | baseline, 6, 9 and 12 months
  BMI will be assessed by measuring height and weight of children

OTHER OUTCOMES:
change in days with asthma symptoms | baseline, 6, 9, 12 months
  days with asthma symptoms will be assessed by parental self-report

CONTACTS AND LOCATIONS:
Overall Officials: Marina Reznik, MD, MS, Principal Investigator — Children's Hospital at Montefiore, Albert Einstein College of Medicine
Locations (1):
- Children's Hospital at Montefiore, Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Walker TJ, Reznik M. In-school asthma management and physical activity: children's perspectives. J Asthma. 2014 Oct;51(8):808-13. doi: 10.3109/02770903.2014.920875. Epub 2014 May 14. PMID 24796650
- [Result] Reznik M, Bauman LJ, Okelo SO, Halterman JS. Asthma identification and medication administration forms in New York City schools. Ann Allergy Asthma Immunol. 2015 Jan;114(1):67-68.e1. doi: 10.1016/j.anai.2014.10.006. Epub 2014 Oct 24. No abstract available. PMID 25454012
- [Result] Jaramillo Y, Reznik M. Do United States' teachers know and adhere to the national guidelines on asthma management in the classroom? A systematic review. ScientificWorldJournal. 2015;2015:624828. doi: 10.1155/2015/624828. Epub 2015 Feb 2. PMID 25729770
- [Result] Kornblit A, Cain A, Bauman LJ, Brown NM, Reznik M. Parental Perspectives of Barriers to Physical Activity in Urban Schoolchildren With Asthma. Acad Pediatr. 2018 Apr;18(3):310-316. doi: 10.1016/j.acap.2017.12.011. Epub 2018 Jan 5. PMID 29309846
- [Result] Cain A, Reznik M. The Principal and Nurse Perspective on Gaps in Asthma Care and Barriers to Physical Activity in New York City Schools: A Qualitative Study. Health Educ Behav. 2018 Jun;45(3):410-422. doi: 10.1177/1090198117736351. Epub 2017 Oct 31. PMID 29084455
- [Result] Reznik M, Islamovic F, Choi J, Leu CS, Rowlands AV. Factors associated with in-school physical activity among urban children with asthma. J Asthma. 2018 May;55(5):492-501. doi: 10.1080/02770903.2017.1340482. Epub 2017 Jul 21. PMID 28696842
- [Result] Cain A, Reznik M. Asthma management in New York City schools: A classroom teacher perspective. J Asthma. 2016 Sep;53(7):744-50. doi: 10.3109/02770903.2015.1135946. Epub 2016 May 17. PMID 27031532
- [Result] Reznik M, Halterman JS. School asthma policies and teachers' confidence and attitudes about their role in asthma management. Ann Allergy Asthma Immunol. 2016 May;116(5):473-5. doi: 10.1016/j.anai.2016.03.005. Epub 2016 Mar 22. No abstract available. PMID 27013055
- [Derived] Reznik M, Islamovic F, Halterman JS, Leu CS, Zhang J, Ozuah PO. Multicomponent intervention for schoolchildren with asthma: Pilot cluster randomized controlled trial. J Allergy Clin Immunol Glob. 2025 Jan 18;4(2):100418. doi: 10.1016/j.jacig.2025.100418. eCollection 2025 May. PMID 40008092
- [Derived] Reznik M, Greenberg E, Cain A, Halterman JS, Ivanna Avalos M. Improving teacher comfort and self-efficacy in asthma management. J Asthma. 2020 Nov;57(11):1237-1243. doi: 10.1080/02770903.2019.1640732. Epub 2019 Jul 17. PMID 31314614